CLINICAL TRIAL: NCT00027911
Title: A Pilot Study of NY-ESO-1 Immunization in Patients With NY-ESO-1/LAGE Antigen Expressing Cancer
Brief Title: Vaccine Therapy and Sargramostim in Treating Patients With Soft Tissue Sarcoma
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Departure of PI
Sponsor: Columbia University (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Purpose: Treatment
Other Study IDs: AAAB2273; CPMC-IRB-13578; LUDWIG-LUD00-024; NCI-G01-2035
Record Dates: First submitted 2001-12-07; First posted 2003-01-27 (Estimated); Last update posted 2013-02-15 (Estimated); Status verified 2013-02

CONDITIONS: Sarcoma
Keywords: adult synovial sarcoma; stage III adult soft tissue sarcoma; recurrent adult soft tissue sarcoma; stage IV adult soft tissue sarcoma; stage II adult soft tissue sarcoma
MeSH Terms: conditions — Sarcoma; Sarcoma, Synovial | interventions — sargramostim

INTERVENTIONS:
Biological: NY-ESO-1 peptide vaccine
Biological: sargramostim

SUMMARY:
RATIONALE: Vaccines may make the body build an immune response to kill tumor cells. Colony-stimulating factors such as sargramostim increase the number of immune cells found in bone marrow or peripheral blood. Combining vaccine therapy with sargramostim may be effective in treating soft tissue sarcoma.

PURPOSE: Phase I trial to study the effectiveness of combining vaccine therapy with sargramostim in treating patients who have stage II, stage III, or stage IV soft tissue sarcoma.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the safety and tolerability of NY-ESO-1 peptide vaccine and sargramostim (GM-CSF) in patients with stage II, III, or IV soft tissue sarcoma expressing NY-ESO-1 or LAGE antigen.
* Determine the immunologic profile (NY-ESO-1 antibody, CD8+ cells, and delayed-type hypersensitivity) in patients treated with this regimen.
* Determine tumor responses in patients treated with this regimen.

OUTLINE: Patients receive NY-ESO-1 peptide vaccine intradermally once every 2 weeks for a total of 6 vaccinations. Patients also receive sargramostim (GM-CSF) subcutaneously once daily beginning 2 days before every vaccination and continuing for 5 days. Treatment continues in the absence of disease progression or unacceptable toxicity.

PROJECTED ACCRUAL: A total of 15 patients will be accrued for this study within 12 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed high-risk stage II, III, or IV soft tissue sarcoma expressing NY-ESO-1 or LAGE antigen (including, but not limited to, synovial sarcoma)
* HLA-A2 allele for NY-ESO-1 peptides
* Declined, failed, or completed standard therapy
* CNS metastases allowed if treated and stable

PATIENT CHARACTERISTICS:

Age:

* 18 and over

Performance status:

* Not specified

Life expectancy:

* At least 3 months

Hematopoietic:

* Hemoglobin at least 9.0 g/dL
* Lymphocyte count at least 500/mm3
* Platelet count at least 100,000/mm3
* No bleeding disorders

Hepatic:

* Bilirubin no greater than 2 mg/dL
* Hepatitis B and C negative

Renal:

* Creatinine no greater than 1.8 mg/dL

Cardiovascular:

* No New York Heart Association class III or IV heart disease

Other:

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* HIV negative
* No other serious illness (e.g., serious infection requiring antibiotics)
* No immunodeficiency disease
* No psychiatric or addictive disorders that would preclude study

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* No prior bone marrow or peripheral blood stem cell transplantation
* At least 4 weeks since prior immunotherapy

Chemotherapy:

* At least 4 weeks since prior chemotherapy (6 weeks for nitrosoureas)
* No concurrent chemotherapy

Endocrine therapy:

* No concurrent steroids except topical or inhaled steroids
* Concurrent noncytotoxic anticancer hormonal therapy allowed (e.g., hormones for breast or prostate cancer)

Radiotherapy:

* At least 4 weeks since prior radiotherapy

Surgery:

* At least 4 weeks since prior surgery

Other:

* At least 4 weeks since prior participation in any other clinical trial involving another investigational agent
* No concurrent antihistamines
* No concurrent non-steroidal anti-inflammatory drugs except low doses for prevention of an acute cardiovascular event or pain control
* No concurrent immunosuppressive agents
* Concurrent noncytotoxic anticancer therapy allowed

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2001-04; Primary Completion 2005-06 (Actual); Study Completion 2005-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kyriakos P. Papadopoulos, MD, Study Chair — Herbert Irving Comprehensive Cancer Center
Locations (1):
- Herbert Irving Comprehensive Cancer Center at Columbia University, New York, New York, United States